CLINICAL TRIAL: NCT01517828
Title: Intranasal Midazolam Versus Intranasal Ketamine to Sedate Newborns for Intubation in Delivery Room.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UF8736; 2011-003216-23 (EudraCT Number)
Record Dates: First submitted 2011-12-12; First posted 2012-01-25 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Respiratory Distress Syndrome; Prematurity of Fetus
Keywords: Intubation; Delivery room; Sedation; Analgesia
MeSH Terms: conditions — Respiratory Distress Syndrome; Agnosia | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine Arm (Experimental): Phial of Ketamine (50mg/5ml) will be used and the dose administered will be 2 mg/kg.
  Interventions: Drug: Sedation by ketamine
- Midazolam Arm (Active Comparator): Phials of midazolam (5mg/5ml)will be used and the dose administered will be 0.2 ml/kg.
  Interventions: Drug: Sedation with Midazolam

INTERVENTIONS:
Drug: Sedation by ketamine — Kétamine (50mg/5ml, Panpharma): for a posology of 2 mg/kg: dose of 0.2 ml/kg Intranasal administration with a 1 ml syringe. Kétamine is a derivated of phencyclidine with a sedative, anesthesic, analgesic and amnesiant activity. Ketamine keeps also a protective reflex of upper respiratory tracts.
  One injection will be done and if after 7 minutes, newborn is not correctly sedated another dose of same product will be done.
  Arms: Ketamine Arm
Drug: Sedation with Midazolam — Midazolam (phyal of 5mg/5ml, Mylan S.A.S.) for a posology of 0.2 mg/kg: dose of 0.2 ml/kg Instillation in intranasal with a syringe of 1 ml. Midazolam is an imidazobenzodiazépine, witj a sedative and hypnotic activity,anxiolytic, anti convulsive and muscle relaxant proprieties.
  One injection will be done and if after 7 minutes, newborn is not correctly sedated another dose of same product will be done.
  Arms: Midazolam Arm

SUMMARY:
Anesthesia is rarely used to intubate newborns in delivery room because of the very difficulty of accessing veins. The investigators hypothesized that intranasal administration of sedative would be an effective alternative. -Midazolam and Ketamine are two drugs used during neonates' intubation. They are also used intranasally in the absence of venous access-In a pilot study the investigators have demonstrated that sedation with Midazolam was effective in 67% of the patients. Efficiency was defined by a specific pain score: FANS < 4 (Faceless Acute Neonatal Pain Scale) and by an impedancemetric Pain monitor < 0.2 spike/s.

The investigators hypothesized that intranasal ketamine would increase procedure effectiveness from 67 to 90%.

* Main objective: To compare newborns sedation quality as they are sedated either by intranasal Midazolam or by intranasal Ketamine during intubation in delivery room.
* Secondary Objectives: To compare intubation quality, hemodynamic and respiratory tolerance, and neurological outcomeat 2 years within the two groups.

DETAILED DESCRIPTION:
Randomized, double blind prospective multicenter study. Patients:-Inclusion criteria: (1) neonates in delivery room (2) Presence of repiratory distress syndrom requiring intubation (Silverman score> 3 and / or FiO2 greater than 30 % in premature infants under 30 weeks and over 40% after 30 weeks (3) hemodynamic stability (mean arterial pressure> 3° percentile)

* Exclusion criteria: (1) Need for intubation in extreme emergency (pneumothorax, meconium aspiration, congenital diaphragmatic hernia, perinatal asphyxia) (2) Birth in the absence of an independent appraiser (3) mother under general anesthesia.
* Number of subjects required: 120 patients (60 per group) over a period of two years. This number was calculated to show a difference in sedation effectiveness from 67 to 90% with an alpha risk of 5% and a beta risk of 20%.
* Study design:

After obtaining parental consent, patients will be randomized in "Midazolam" arm or in "Ketamine" arm . Midazolam (0.2mg/kg = 0.2ml/kg) or Ketamine (2mg/kg = 0.2 ml/kg) are instilled in the nose, using a 1 ml syringe. The gesture will be directed by a physician having yet successfully completed a minimum of 50 intubations. After sedation completion, intubation decision will be taken at the onset of muscle relaxation or on the occurrence of apnea.

* The clinical pain score will be evaluated on film a posteriori by two independent observers using a scale of hetero pain assessment.-Pain will be evaluated through the study of skin conductance.
* The quality of intubation will be judged by the number of attempts required and by the duration of glottis exposure.
* Hemodynamic and respiratory tolerances will be judged by measuring respectively variations in blood pressure, heart rate, FiO2 and the oxygen saturation.

The neurological follow-up will be carried out according to Brunet-Lezine developmental scale at the age of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Neonates in delivery room
* Presence of respiratory distress syndrom requiring intubation (Silverman score> 3 and / or FiO2 greater than 30 % in premature infants under 30 weeks and over 40% after 30 weeks
* Hemodynamic stability (mean arterial pressure> 3° percentile)

Exclusion Criteria:

* Need for intubation in extreme emergency (pneumothorax, meconium aspiration, congenital diaphragmatic hernia, perinatal asphyxia)
* Birth in the absence of an independent appraiser
* Mother under general anesthesia

Max Age: 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Newborns sedation quality | during the 10 minutes of intubation
  The sedation quality of 2 newborns groups will be compared during the 10 minutes of intubation directly in delivery room and after on the film Pain evaluation done by a Specific clinical Score : the Faceless Acute Neonatal pain Scale (FANS) noted by two independent professional persons. And for Montpellier center, evaluation of pain by cutaneous conductance

SECONDARY OUTCOMES:
intubation quality | during the 10 minutes of intubation
  Intubation quality will be evaluated and compared between the two groups by numbers of attempts, duration of glottis exposition (from introduction to withdrawal of laryngoscop)
hemodynamic and respiratory tolerance | during 24 hours after intubation
  Hemodynamic tolerance will be measured by Mean Arterial Pressure every 3 minutes before and after product instillation and during the intubation. After intubation, measure of Mean Arterial Pressure will be done every 10 minutes during 1 hour and after every hour until 24 hours. Cardiac frequency and cardiac fraquency variations will be measured and analyzed.
  Respiratory tolerance will be evaluated by continuing measure of SpO2, delay of instillation of surfactant dose and the need to administer un second dose of surfactant
neurological outcome at 2 years within the 2 groups | 2 years after the treatment
  Prevalence of neurological complications (intraventricular hemorragies, periventricular leucomalacies), development quotient at 2 years (Brunet Lezine scale)will be evaluated and compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Christophe CM MILESI, MD, Principal Investigator — University Hospital, Montpellier
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire, Montpellier
  - Centre Hospitalier Universitaire, Nîmes
  - Centre Hospitalier Général, Perpignan

REFERENCES:
- [Derived] Milesi C, Baleine J, Mura T, Benito-Castro F, Ferragu F, Thiriez G, Thevenot P, Combes C, Carbajal R, Cambonie G. Nasal midazolam vs ketamine for neonatal intubation in the delivery room: a randomised trial. Arch Dis Child Fetal Neonatal Ed. 2018 May;103(3):F221-F226. doi: 10.1136/archdischild-2017-312808. Epub 2017 Aug 17. PMID 28818854